CLINICAL TRIAL: NCT07371351
Title: The Effect of EMST and Triflo Devices on Acoustic and Aerodynamic Parameters of Sound and Sound Fatigue in Academics: A Randomized Controlled Study
Brief Title: "Effects of EMST and Triflo on Voice Parameters and Vocal Fatigue"
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Eda Uzuner, lecturer, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IMU-DKT-EU-01
Record Dates: First submitted 2025-12-23; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Voice Fatigue; Voice Disorder; Academic Voice Use and Voice Fatigue; Academician's Risk of Developing Voice Disorder; Voice Disorder Prevention in Academics
Keywords: Voice Disorders; Vocal Fatigue; Professional Voice Users; Respiratory Muscle Training; Acoustic Analysis
MeSH Terms: conditions — Voice Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial. This is a randomized controlled trial. The study will consist of two groups: Group 1 will receive only EMST, Group 2 will receive both EMST and Triflo, Group 3 will receive Triflo, and Group 4 will be the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- first experimental group (Experimental): triflo will be applied
  Interventions: Device: Triflo
- second experimental groups (Experimental): EMST application will be performed.
  Interventions: Device: EMST
- third experimental groups (Experimental): EMST and Triflo applications will be carried out.
  Interventions: Device: Triflo; Device: EMST
- control groups (No Intervention)

INTERVENTIONS:
Device: Triflo — The TriFlo Breathing Exercise Device is scientifically designed to assist in performing breathing exercises that may be prescribed by doctors. This device increases participants' breath volume. Participants hold the device upright by its plastic parts and try to lift the balls upwards while inhaling. Alternatively, participants can invert the device by holding the plastic parts (the balls will fall down) and try to lift the balls upwards while exhaling. Participants will be asked to perform this exercise 5 days a week, 4 hours a day, in 3 sets of 10 exhalations and 10 inhalations.
  Arms: first experimental group; third experimental groups
Device: EMST — EMST is a rehabilitation approach that uses a device to increase and activate the maximum pressure of the respiratory muscles. These muscles are important for powerful exhalation, coughing, and swallowing. EMST Week 1 Exercise Steps
  a. The participant is instructed to place the nasal plug on their nasal bone. b. The participant is asked to take a deep breath and not exhale.
  c. The participant is instructed to place the mouthpiece behind their teeth, inside their mouth, and press their lips firmly against the mouthpiece, pressing down on the sides of their cheeks if necessary.
  d. Participants are instructed to exhale forcefully and quickly, using their chest and abdominal muscles to push the air through the device. This exhalation effort should only take a few seconds for the air to pass.
  e. Participants are instructed to rest for at least 15-30 seconds, and to rest between breaths as well. The muscles need time to prepare for the next set.
  f. Participants repeat this exercise 5 times
  Arms: second experimental groups; third experimental groups

SUMMARY:
A healthy voice is essential for meeting professional and communicative demands, particularly for professional voice users such as academics, who are at increased risk of voice disorders due to prolonged and intensive voice use, unfavorable acoustic conditions, and stress. Voice disorders often result from inadequate respiratory support, leading to compensatory laryngeal overuse, vocal fatigue, and deterioration in voice quality. Although traditional voice therapy emphasizes diaphragmatic breathing, it does not enhance respiratory capacity because it lacks resistance. This study aims to investigate the effects of resistance-based breathing exercises using the Expiratory Muscle Strength Trainer (EMST 150) and triflo devices on respiratory capacity, acoustic and aerodynamic voice parameters, and vocal fatigue in academics. The findings are expected to contribute to the literature and support the use of EMST as a preventive and therapeutic approach for occupational groups at risk of voice disorders.

DETAILED DESCRIPTION:
A healthy voice should provide information about a person's age, gender, and emotional state, while also meeting their professional, social, and communicative needs. A voice disorder is generally a change in voice quality, pitch, and/or loudness that differs from what is expected for someone of the same age or gender. In the presence of a voice disorder, the voice does not represent the speaker and cannot meet their professional, social, and communicative needs. There are many risk factors that cause voice disorders. One of these is occupation.

Speaking excessively long and loudly or at a high pitch due to one's profession is defined as voice misuse and can cause voice disorders. For example, members of professions that require intensive and prolonged use of their voices (teachers, imams, academics, telephone operators, lawyers, theater actors) are more likely to experience voice disorders. Individuals who use their voices as a primary means of communication while performing their professions are defined as professional voice users.

Although professional voice users from different occupational groups may seem to fall under the same heading, they differ in various aspects such as the frequency and method of voice use. This differentiation was classified into four levels of voice by Koufman and Isaacson (1991), and academics were included in the category of professional voice users. Voice disorders are seen in 10% of the general population and 50% of professional voice users. Despite this, there is an insufficient number of studies examining the prevalence of voice disorders in academics, risk factors, and research aimed at evaluating, diagnosing, and preventing observed voice disorders.

Professional voice users have to use their voices more effectively and intensely due to their intensive voice use, and this leads to a need for a stronger and healthier voice compared to other individuals. Risk factors that cause voice disorders in teachers, such as speaking loudly for long periods, noisy and acoustically poor working environments, dry and dusty air, and stress, also apply to academics.

In professions with high voice demands, such as teaching and academia, in addition to reducing or eliminating voice-related problems, preventive intervention programs should be implemented, and the voice should be strengthened to make it resistant to long-term and intensive use. Voice enhancement and long-term use are highly related to respiration, a component of the voice production mechanism.

Respiration, in addition to ventilating the body, provides the exhaled airflow that forms the basis of all voice and speech production. Two aspects of respiration that directly affect voice production are breath support and breath control. Breath support refers to the stabilization of body structures to create adequate air pressure and airflow; breath control refers to how an individual regulates and coordinates airflow for all activities, including speech. Difficulty in establishing and/or maintaining breath support and breath control, such as difficulties in inhaling and/or exhaling air or obtaining sufficient air, can negatively affect voice production. For example, if the respiratory system cannot provide sufficient breath support for voice production, the laryngeal system may overcompensate, leading to voice fatigue, tissue changes in the vocal cords, and changes in voice quality.

Therefore, respiratory support plays an important role in the prevention and rehabilitation of voice disorders. However, changing an individual's type of respiration (clavicular, chest, diaphragmatic) and capacity is not easy or quick. Current voice therapy approaches necessarily include breathing, but they are based on teaching diaphragmatic breathing. Teaching diaphragmatic breathing allows individuals to utilize their existing respiratory capacity, but the absence of resistance does not increase respiratory capacity. This study aims to improve the respiratory capacity and voice quality of academics who require long-term voice production, while reducing vocal fatigue, using an EMST device that enables breathing exercises against resistance. To this end, breathing exercises will be performed using the Expiratory Muscle Strength Trainer (EMST 150) and triflo devices, which allow for pressure adjustment. The application of the EMST device in academics at risk of voice disorders and the results will provide data for the literature. If the study shows an increase in acoustic voice quality, aerodynamic parameters, and exhaled volume, and a decrease in vocal fatigue, the EMST device can be included in therapy for occupational groups with or at risk of voice disorders.

ELIGIBILITY:
Inclusion Criteria:

Having taught for at least 2 academic semesters as an academic. Having taught at least 9 hours of face-to-face classes per week. Not having been diagnosed with an organic voice disorder. Not smoking. Not being in a menstrual cycle during the pre-, mid- and post-tests.

Exclusion Criteria:

Being Pregnancy, hypertension disease have a history of stroke, heart anomaly disease chronic asthma disease emphysema or obstructive pulmonary disease, have a any surgery in the skull base and neck region, have a any neurogenic or psychological diagnosis or condition.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Measurement of vocal fatigue | The study will continue for 4 months from the start of the study.
  To assess vocal fatigue, participants will complete a vocal fatigue scale before starting the exercises. Participants will fill out this scale themselves. They will rate the parameters related to vocal fatigue on a scale of 0 to 4. Higher scores indicate greater fatigue. The validity and reliability of the vocal fatigue scale have been established in Turkish. Participants will be asked to complete this scale again in the 3rd week of the exercises and again in the 5th week, which is the final week of the exercises. They will also be asked to complete it again 2 months after the completion of the exercises for follow-up.
measurement of acoustic parameters of voice | The study will continue for 4 months from the start of the study.
  In acoustic measurement, participants will have their measurements taken before starting the exercises.For acoustic parameters of the voice, jitter, shimmer, noise-harmonic ratio, and harmonic-noise ratio parameters will be measured by recording via the Multi-Dimensional Voice Program (MDVP). Furthermore, for acoustic parameters of the voice, the extra smooth cepstral peak prominence value and the Acoustic Voice Quality Index (AVQI) score will be calculated using Praat. These measurements will be repeated 3 weeks after the start of exercises, 5 weeks after the completion of exercises, and 2 months after the completion of exercises during follow-up.
Aerodynamic measurement of the voice, | The study will continue for 4 months from the start of the study.
  For the aerodynamic measurement of voice, participants will be asked to produce the sounds /s/ (measuring lung capacity), /z/ (vocal cord closure time), and /a/ (average sound production time), and the duration will be recorded. An s/z ratio close to 1 or between 1 and 1.3 is considered normal. For /a/ phonation, a normal adult is expected to produce sounds of 27-28 seconds. Participants' values will be recorded before the exercise, at the 3rd week of exercise, at the 5th week after the exercise, and again at 2 months post-exercise for follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: eda Uzuner, phd candidate, Study Director — Medipol University
Locations (1):
- İstanbul Medipol Üniversitesi- MEDKOM, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No